CLINICAL TRIAL: NCT06656481
Title: COMPARISON OF PHOENIXIN-14 LEVELS IN UMBILICAL CORD BLOOD ACCORDING TO BIRTH WEIGHT IN TERM INFANTS: ARE PHOENIXIN-14 LEVELS LINKED TO BIRTH WEIGHT AND MATERNAL DIABETES?
Brief Title: Comparison of Phoenixin-14 Levels in Term Babies
Acronym: PNX-14
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, RAMAZAN KEÇECİ, NEONATOLOGIST, MD, PRINCIPAL INVESTIGATOR, Konya City Hospital
Other Study IDs: 2022/005
Record Dates: First submitted 2024-10-19; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Diabetes, Gestational; Weight, Fetal
Keywords: newborn; phoenixin-14; birthweight
MeSH Terms: conditions — Diabetes, Gestational; Fetal Weight; Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1. Small for Gestational Age Babies (SGA): Infants with birth weight below the 10th percentile are classified as small for gestational age (SGA
- 2. Large for Gestational Age Babies (LGA): infants above the 90th percentile are classified as large for gestational age (LGA)
- 3. Appropriate for Gestational Age Babies (AGA): between the 10th and 90th percentiles are classified as appropriate for gestational age
- 4. GDM: babies of Mothers with gestational diabetes mellitus

SUMMARY:
INTRODUCTION Birth weight and pregnancy week are determinants of mortality and morbidity of newborn infants. Birth weights by gestational week are associated with accompanying diseases in the later stages of life (1). Infants with a birth weight below the 10th percentile by gestational week are defined as small for gestational age (SGA), those with a birth weight above the 90th percentile are defined as large for gestational age (LGA), and those with a birth weight between the 10th and 90th percentiles are defined as appropriate for gestational age (AGA) (2). In LGA and SGA infants, problems such as hypoglycemia, hypoxia, polycythemia, and respiratory support may be encountered in the neonatal period. These infants may also experience diseases that affect the quality and duration of life at later ages, such as metabolic syndrome, obesity, cardiovascular diseases, and diabetes mellitus (1, 2). Gestational diabetes mellitus (GDM) is the most common complication during pregnancy and is defined as any degree of glucose intolerance that begins or is first recognized during pregnancy (3). GDM has long been associated with obstetric and neonatal complications, particularly those related to high birth weight, and is increasingly recognized as a risk factor for future cardiometabolic disease in the child. As the causes of serious health problems can be attributed to maternal illness or changes in birth weight, these issues continue to be investigated (4).

Phoenixin (PNX) is a neuropeptide first described by Yosten et al. in 2013 (5). The most common isoforms of PNX, phoenixin-14 (PNX-14) and phoenixin-20 (PNX-20), exhibit similar biological activities and are peptides composed of 14 and 20 amino acids, respectively (5). In the initial characterization of PNX, it was reported to be crucial for normal reproductive function through its effects on the hypothalamus-pituitary-gonadal axis. The literature provides further evidence for the role of PNX in reproductive functions and suggests that it also plays a role in other aspects of brain-mediated and peripheral physiology. In addition, there is some evidence demonstrating that PNX affects the heart, diet, memory, and anxiety (6). Animal studies of PNX-14 have shown that PNX-14 has an important role in the central control of feeding behavior and metabolic homeostasis. In addition to correlations between PNX-14 and body mass index (BMI), studies have shown that PNX-14 modulates food intake and feeding behavior (7). PNX-14 is a neuropeptide known to prevent oxidative damage and stimulate insulin secretion. Animal studies have shown that PNX-14 treatments prevent pancreatic damage and β-cell loss by reducing oxidative stress (8). A study indicating that PNX-14 plays an important role in the occurrence of diabetes and obesity found that PNX-14 concentrations were significantly lower in patients with type 2 diabetes mellitus than in healthy individuals (9, 10).

In this study, we investigated the relationships between normal (AGA), low (SGA), and high (LGA) birth weight according to gestational week of pregnancy and phoenixin-14 levels in the umbilical cord blood of healthy infants of healthy mothers and infants of mothers diagnosed with GDM regardless of birth weight.

DETAILED DESCRIPTION:
INTRODUCTION Birth weight and pregnancy week are determinants of mortality and morbidity of newborn infants. Birth weights by gestational week are associated with accompanying diseases in the later stages of life (1). Infants with a birth weight below the 10th percentile by gestational week are defined as small for gestational age (SGA), those with a birth weight above the 90th percentile are defined as large for gestational age (LGA), and those with a birth weight between the 10th and 90th percentiles are defined as appropriate for gestational age (AGA) (2). In LGA and SGA infants, problems such as hypoglycemia, hypoxia, polycythemia, and respiratory support may be encountered in the neonatal period. These infants may also experience diseases that affect the quality and duration of life at later ages, such as metabolic syndrome, obesity, cardiovascular diseases, and diabetes mellitus (1, 2). Gestational diabetes mellitus (GDM) is the most common complication during pregnancy and is defined as any degree of glucose intolerance that begins or is first recognized during pregnancy (3). GDM has long been associated with obstetric and neonatal complications, particularly those related to high birth weight, and is increasingly recognized as a risk factor for future cardiometabolic disease in the child. As the causes of serious health problems can be attributed to maternal illness or changes in birth weight, these issues continue to be investigated (4).

Phoenixin (PNX) is a neuropeptide first described by Yosten et al. in 2013 (5). The most common isoforms of PNX, phoenixin-14 (PNX-14) and phoenixin-20 (PNX-20), exhibit similar biological activities and are peptides composed of 14 and 20 amino acids, respectively (5). In the initial characterization of PNX, it was reported to be crucial for normal reproductive function through its effects on the hypothalamus-pituitary-gonadal axis. The literature provides further evidence for the role of PNX in reproductive functions and suggests that it also plays a role in other aspects of brain-mediated and peripheral physiology. In addition, there is some evidence demonstrating that PNX affects the heart, diet, memory, and anxiety (6). Animal studies of PNX-14 have shown that PNX-14 has an important role in the central control of feeding behavior and metabolic homeostasis. In addition to correlations between PNX-14 and body mass index (BMI), studies have shown that PNX-14 modulates food intake and feeding behavior (7). PNX-14 is a neuropeptide known to prevent oxidative damage and stimulate insulin secretion. Animal studies have shown that PNX-14 treatments prevent pancreatic damage and β-cell loss by reducing oxidative stress (8). A study indicating that PNX-14 plays an important role in the occurrence of diabetes and obesity found that PNX-14 concentrations were significantly lower in patients with type 2 diabetes mellitus than in healthy individuals (9, 10).

In this study, we investigated the relationships between normal (AGA), low (SGA), and high (LGA) birth weight according to gestational week of pregnancy and phoenixin-14 levels in the umbilical cord blood of healthy infants of healthy mothers and infants of mothers diagnosed with GDM regardless of birth weight.

MATERIALS AND METHODS We obtained approval for this prospective study from the Karatay University Ethics Committee (Ethics Committee Decision No: 2022/005) and Konya City Hospital. We conducted the research between December 2022 and April 2024 at Konya City Hospital in the Department of Obstetrics and Gynecology, the Neonatal Intensive Care Unit, and the Department of Medical Biochemistry (Clinical Trials ID: NCT).

Patients Infants with multiple congenital anomalies, chorioamnionitis, and preeclampsia; infants who were born after premature rupture of membranes; infants who needed intensive care; and otherwise ill or premature infants were excluded from the study. Infants whose mothers had any disease other than diabetes were also excluded. Healthy term infants (born between 370/7 and 426/7 weeks) born by spontaneous vaginal delivery or cesarean section were included in the study. The demographic and neonatal data and the PNX-14 levels of the patients included in the study were recorded.

The sample size was determined with two-way independent-samples t-test power analysis based on previous studies. According to previous similar studies, phoenixin-14 ratios with an error margin of 0.05, actual power level of 0.9554213, and effect size of 1.41 would require a minimum of 24 deliveries (12 vaginal deliveries and 12 cesarean sections) for each pairwise comparison; however, aiming to reduce the margin of error, we planned to include 40 infants in each group. Four different groups were considered in this study:

1. Infants with low birth weight by gestational week (SGA): Of the 42 infants in this group whose mothers agreed to participate in the study, 2 were excluded due to incomplete laboratory data or hospitalization in the neonatal intensive care unit due to sepsis, and 40 SGA infants (20 born by spontaneous vaginal delivery and 20 by cesarean delivery) were included in the study.
2. Infants with normal birth weight by gestational week (AGA): Of the 47 infants in this group, 7 were excluded due to incomplete laboratory data or mothers declining to participate, and 40 AGA infants (20 born by spontaneous vaginal delivery and 20 by cesarean delivery) were included in the study.
3. Infants with high birth weight by gestational week (LGA): Of the 44 babies in this group whose mothers agreed to participate in the study, 4 were excluded due to suspected sepsis, incomplete laboratory data, or neonatal intensive care unit hospitalization, and 40 LGA infants (20 born by spontaneous vaginal delivery and 20 by cesarean delivery) were included in the study.
4. Infants whose mothers had gestational diabetes mellitus (GDM): Of the 41 infants in this group whose mothers agreed to participate in the study, 1 was excluded due to missing antenatal demographic data, and 40 infants (4 born by spontaneous vaginal delivery and 36 by cesarean delivery) were included in the study.

Biochemical analysis After obtaining informed consent from their parents, umbilical cord blood samples were collected from all infants. The obtained blood samples were centrifuged within 6 hours and the serum was separated. Following the manufacturer's instructions, commercial kits (BT Lab Bioassay Technology Laboratory Human ELISA Kits, Shanghai Korain Biotech, Shanghai, China) were used to perform enzyme immunoassay analyses of serum PNX-14 levels. Using an ELx800 Absorbance Microplate Reader (Biotech, Winooski, VT, USA), the absorbance was measured at 450 nm. The concentration values for PNX-14 were expressed in ng/L. The kit's sensitivity was 8.19 ng/L and the standard curve range was 20-3800 ng/L. Interassay and intraassay differences were less than 10% and 8%, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants (born between 37+0 and 42+6 weeks) delivered by spontaneous vaginal delivery or cesarean section were included in the study

Exclusion Criteria:

* Infants with multiple congenital anomalies
* Chorioamnionitis
* Preeclampsia
* Mothers had premature rupture of membranes,
* Requiring intensive care unit

Ages: 1 Minute to 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1. Small for Gestational Age Babies (SGA): (20 spontaneous vaginal births, 20 cesarean births).
  2. Appropriate for Gestational Age Babies (AGA): (20 spontaneous vaginal births, 20 cesarean births).
  3. Large for Gestational Age Babies (LGA): (20 spontaneous vaginal births, 20 cesarean births).
  4. Babies of Mothers with Gestational Diabetes Mellitus (GDM): 4 spontaneous vaginal births, 36 cesarean births).
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
COMPARISON OF CORD BLOOD PHOENIXIN-14 LEVELS ACCORDING TO BIRTH WEIGHTS IN TERM INFANTS | between December 2022 and April 2024.
  In our study, we investigated the relationship between the cord blood levels of phoenixin-14 and the birth weights of healthy term infants born to healthy mothers, classified as normal (AGA), low (SGA), or high (LGA) based on gestational age, as well as mothers diagnosed with gestational diabetes mellitus (GDM) regardless of birth weight.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Keçeci, Principal Investigator — Konya City Hospital; beyza özcan, specialist, Study Chair — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
PROTOCOL CAN BE SHARED WHEN THE STUDY IS PUBLISHED
Supporting Information: Study Protocol

REFERENCES:
- See also: PUBMED — https://pubmed.ncbi.nlm.nih.gov/